CLINICAL TRIAL: NCT04681040
Title: Monitoring of COVID-19 Using Urine POC Kit
Brief Title: Risk Stratification of COVID-19 Using Urine Biomarkers
Status: Active, not recruiting | Type: Observational
Sponsor: National Center for Global Health and Medicine, Japan (Other Government)
Responsible Party: Principal Investigator, Eisei Noiri, MD, PhD, FASN, Director General, National Center Biobank Network, National Center for Global Health and Medicine, Japan
Other Study IDs: NCGM-G-003654-00; 20he0822003j0001 (Other Grant/Funding Number: AMED)
Record Dates: First submitted 2020-12-19; First posted 2020-12-23 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Covid19; Urine; Biomarker; Acute Respiratory Failure With Hypoxia
Keywords: L-type Fatty Acid-binding Protein, beta 2 microglobulin
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Serum and plasma biomarkers of inflammation / cytokine storm, coagulation, and ischemia / organ injury.
  2. Urine L-FABP, Urine beta2 microgloburin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UrBMC19 Group (International Cooperative Group): The examination of urine for mild pre-diagnosed COVID-19 cases are conducted to evaluate the risk classification and detect the effectiveness of early intervention by COVID-19 treatment such as dexamethasone, chloroquine, remdesivir, ivermectin, actemra, and so forth within the period of 14 days after starting the intervention.

SUMMARY:
Coronavirus disease 2019 (COVID-19) is caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and in infected patients, it produces symptoms which range from completely asymptomatic to those expressing severe illness. Early recognition of those developing severe manifestations allows for rapid and appropriate intervention, including admission to intensive care unit and intensive care therapy, such as mechanical ventilation. A current problem is that only limited data exist predicting the clinical course of COVID-19. This study will determine whether non-invasive urinalysis is useful in assessing and predicting the severity or clinical course of patients with COVID-19.

DETAILED DESCRIPTION:
This study will conduct to elucidate the following clinical question;

1. if the single urinary biomarker or the combination of urinary biomarkers will clarify the risk of COVID-19 confirmed mild cases. These biomarkers must be warranted to clinical use based on the evaluation by either CE or PMDA or FDA. Examination should be done within 72 h after the start of COVID-19.
2. if above addressed biomarker can classify the effectiveness of therapy directed to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 confirmed cases by qPCR exam or equivalent.
* Those who agreed to join this study
* Those who received treatment at NCGM, affiliated hospital and institute including accommodation facilities for observational purposes.

Exclusion Criteria:

* Age less than 20
* Those who do not have smart phone (no personal contract)
* eGFR less than 30
* Any pre-existing illness with fever, weakness, or respiratory difficulties, Pregnancy or breastfeeding.
* Doctors' judgements to inappropriate for inclusion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 confirmed case without severe symptoms.
Sampling Method: Probability Sample
Enrollment: 964 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-03-25 (Estimated)

PRIMARY OUTCOMES:
Risk Stratification of COVID-19 Participants Using Urine Biomarkers | 10 days after starting the initial examination.
  Urine L-FABP will be measured to detect the risk in COVID-19 confirmed cases focusing to no symptom, mild case, and moderate case. Urine beta2 microglobulin will be measured to detect the risk in COVID-19 confirmed cases. Urine L-FABP and beta2 microgloburin will be combined to examine the improvement on risk classification. The risk to develop hypoxic condition, adopted from NEJM 382:1787, 2020 (PMID: 32187464), will be pre-determined by single or dual urine biomarkers using definite cut-off values.
Prediction of COVID-19 Treatment by Urine L-FABP | 14 days after starting the initial intervention.
  The treatment efficacy of a certain specific treatment (ex. dexamethasone, tocilizumab, remdesivir, ivermectin, favipiravir, Hydroxychloroquine, etc) to COVID-19 will be predicted through the initial urine L-FABP level in mild to moderate cases.

SECONDARY OUTCOMES:
Increase of O2 support, hospital days, worsening of chest X-ray and CT, and survival rate, at 14 and/or 30 days. | 30 days after starting the initial examination.
  Applicability of urine L-FABP and beta2 microgloburin will be measured. Single urine biomarker (L-FABP or beta2 microgloburin) or those combination will be evaluated for predictions such as; i) increase of O2 & respiratory supports, ii) increase of hospital days, iii) worsening level of chest X-ray & CT, and iv) survival rate and SOFA in ICU. At 14 and/or 30 days after the inclusion these clinical parameters will be evaluated based on the cut off value of single urine biomarker (L-FABP or beta2 microgloburin) and those aggregates.
Comparison of Risk Stratification with Other Biomarkers | 7 days and 10 days after starting the initial examination.
  Urine L-FABP and beta2 microgloburin will be measured. Single urine biomarker (L-FABP or beta2 microgloburin) or those combination will be compared with d-Dimer and IL-6 for the risk evaluation of COVID-19 in te scope of Outcome 3.

CONTACTS AND LOCATIONS:
Overall Officials: Eisei Noiri, M.D., Ph.D., Principal Investigator — National Center for Global Health and Medicine
Locations (7):
- MD Mount Sinai, Baltimore, Maryland, United States
- Hospital das Clinicas Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil
- Danish National Biobank, Copenhagen, Denmark
- Japan (3):
  - Shonan General Hospital, Kamakura, Kanagawa
  - National Center Global Health and Medicine, Shinjuku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
- Unilab Group, Manila, Philippines

REFERENCES:
- [Background] Katagiri D, Ishikane M, Asai Y, Kinoshita N, Ota M, Moriyama Y, Ide S, Nakamura K, Nakamoto T, Nomoto H, Akiyama Y, Miyazato Y, Suzuki T, Okuhama A, Kanda K, Wakimoto Y, Morioka S, Saito S, Yamamoto K, Ujiie M, Hayakawa K, Kustuna S, Yanagawa Y, Terada J, Takasaki J, Izumi S, Hojo M, Hinoshita F, Sugiyama M, Noiri E, Mizokami M, Ohmagari N, Sugiyama H. Evaluation of Coronavirus Disease 2019 Severity Using Urine Biomarkers. Crit Care Explor. 2020 Jul 31;2(8):e0170. doi: 10.1097/CCE.0000000000000170. eCollection 2020 Aug. PMID 32766565
- [Background] Noiri E, Doi K, Negishi K, Tanaka T, Hamasaki Y, Fujita T, Portilla D, Sugaya T. Urinary fatty acid-binding protein 1: an early predictive biomarker of kidney injury. Am J Physiol Renal Physiol. 2009 Apr;296(4):F669-79. doi: 10.1152/ajprenal.90513.2008. Epub 2008 Nov 19. PMID 19019918
- [Background] Yamamoto T, Noiri E, Ono Y, Doi K, Negishi K, Kamijo A, Kimura K, Fujita T, Kinukawa T, Taniguchi H, Nakamura K, Goto M, Shinozaki N, Ohshima S, Sugaya T. Renal L-type fatty acid--binding protein in acute ischemic injury. J Am Soc Nephrol. 2007 Nov;18(11):2894-902. doi: 10.1681/ASN.2007010097. Epub 2007 Oct 17. PMID 17942962
- [Background] Doi K, Noiri E, Sugaya T. Urinary L-type fatty acid-binding protein as a new renal biomarker in critical care. Curr Opin Crit Care. 2010 Dec;16(6):545-9. doi: 10.1097/MCC.0b013e32833e2fa4. PMID 20736829
- [Background] Tantry US, Bliden KP, Cho A, Walia N, Dahlen JR, Ens G, Traianova M, Jerjian C, Usman A, Gurbel PA. First Experience Addressing the Prognostic Utility of Novel Urinary Biomarkers in Patients With COVID-19. Open Forum Infect Dis. 2021 May 26;8(7):ofab274. doi: 10.1093/ofid/ofab274. eCollection 2021 Jul. PMID 34250193
- [Background] Katagiri D, Asai Y, Ohmagari N, Ishikane M, Hikida S, Iwamoto N, Nagashima M, Suzuki M, Takano H, Takasaki J, Hojo M, Sugiyama H, Tokunaga K, Miyashita Y, Omata M, Ohata K, Bliden KP, Tantry US, Dahlen JR, Sugaya T, Gurbel PA, Noiri E. Urinary L-Type Fatty Acid-Binding Protein Predicts Oxygen Demand of COVID-19 in Initially Mild Cases. Crit Care Explor. 2023 Mar 9;5(3):e0873. doi: 10.1097/CCE.0000000000000873. eCollection 2023 Mar. PMID 36910457
- [Background] Noiri E, Katagiri D, Asai Y, Sugaya T, Tokunaga K. Urine oxygenation predicts COVID-19 risk. Clin Exp Nephrol. 2024 Jul;28(7):608-616. doi: 10.1007/s10157-023-02456-5. Epub 2024 Feb 24. PMID 38400935